CLINICAL TRIAL: NCT02169531
Title: Pilot Study of a Cell-Based Therapy for Treatment of Hyperglycemia in Type 2 Diabetes Mellitus
Brief Title: Ex Vivo Immunotherapy for Hyperglycemia in Type 2 Diabetes Mellitus
Acronym: DISC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: B & Y Technologies (Industry)
Collaborators: Guangzhou No.12 People's Hospital (Other Government); The 12th People's Hospital of Shenzhen City (Unknown)
Responsible Party: Principal Investigator, Demao Yang, Chief Scientist, B & Y Technologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DISCOVER 1
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus; Hyperglycemia
Keywords: Diabetes Mellitus Type 2; Hyperglycemia; Immunotherapy; Autologous
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ex vivo activated immune cells (Experimental): Up to 20 patients diagnosed with type 2 diabetes mellitus and hyperglycemia will be enrolled and assigned to a single treatment group. Patients will give a small amount of peripheral blood and the blood will be processed and cultured in our laboratory. The ex vivo activated autologous blood cells will be infused intravenously back to patients. The treatment will be done twice a week for consecutive 4 weeks. The metabolic parameters of patients before and after the therapy will be compared to determine if the therapy is safe and effective.
  Interventions: Drug: ex vivo Activated Immune Cells

INTERVENTIONS:
Drug: ex vivo Activated Immune Cells — The patients who take medication before the enrollment will be required to reduce at least half the amount of the medication before the treatment. The reduction of the medication will continue during and after the therapy until the levels of plasma hemoglobin A1c (HbA1c) increase to equal or above the levels of the baseline measured before the treatment.

SUMMARY:
Diabetes mellitus type 2 is a long-term metabolic disorder that is primarily characterized by insulin resistance, relative insulin deficiency and hyperglycemia. Our hypotheses is that liver would be the primary organ responsible for the metabolic disorder because of some unknown defects, where sugar would not be efficiently converted to glycogen and fat, leading to hyperglycemia. The constant hyperglycemia would keep pressure on beta-cells in the pancreas to eventually exhaust their ability to produce and secret sufficient amount of insulin, exacerbating the disease. The Immunotherapy would enhance the liver functions and correct the abnormal sugar metabolism. In addition, the ex vivo activated cells produce and secret growth factors which would help endothelial cells of blood vessels to reproduce and grow, resulting in reduced arteriosclerosis.

DETAILED DESCRIPTION:
We plan to recruit 20 patients with type 2 diabetes mellitus who suffer hyperglycemia with or without medication. The patients will come to our hospitals for the treatment. A small amount of peripheral blood will be drawn and processed and cultured in our laboratory. The cultured cells (autologous) will be infused intravenously back to patients. Levels of plasma hemoglobin A1c (HbA1c) and other metabolic parameters before and after the therapy will be compared. The therapy is planned to take four weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with type 2 diabetes mellitus.
* 2. 25 years of age or older. Both sexes.
* 3. HbA1c ≧6.5% for more than 6 months with or without medication.
* 4. Capability of providing informed consent.

Exclusion Criteria:

* 1. History of malignancy.
* 2. Patients with active infections.
* 3. Seropositivity for HIV infection.
* 4. History of myocardial infarction or unstable angina in the previous 3 months.
* 5. Pregnancy or nursing.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Hemoglobin A1c (HbA1c) at up to 27 weeks. | Point 1: The week (week 1) before the first cell infusion assessed as the baseline; Point 2: The week (week 6) after the last cell infusion; Point 3 and after: every 4 weeks up to 27 weeks.

SECONDARY OUTCOMES:
Change from Baseline Lipid Profile at up to 27 weeks. | Point 1: The week (week 1) before the first cell infusion assessed as the baseline; Point 2: The week (week 6) after the last cell infusion; Point 3 and after: every 4 weeks up to 27 weeks.
  Lipid profile includes cholesterol, triglycerides, HDL cholesterol and LDL cholesterol.

OTHER OUTCOMES:
Change from Baseline Symptoms at up to 27 weeks. | Point 1: The week (week 1) before the first cell infusion assessed as the baseline; Point 2: The week (week 6) after the last cell infusion; Point 3 and after: every 4 weeks up to 27 weeks.
  The symptoms include insomnia, anorexia, fatigue, frequent trips to the bathroom, unquenchable thirst and blurred vision.

CONTACTS AND LOCATIONS:
Overall Officials: Lingzhen Chen, MD, Principal Investigator — The 12th People's Hospital of Guangzhou.
Locations (2):
- China (2):
  - The 12th People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The 12th People's Hospital of Shenzhen, Shenzhen, Guangdong